CLINICAL TRIAL: NCT04274101
Title: Nifurtimox Versus Benznidazole Effectiveness and Tolerance for Chagas Disease Treatment, Retrospective Cohort
Brief Title: Nifurtimox Versus Benznidazole Effectiveness and Tolerance for Chagas Disease Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Responsible Party: Principal Investigator, Dr Jaime Altcheh, PHD MD, Hospital de Niños R. Gutierrez de Buenos Aires
Other Study IDs: Nifurtimox vs. Benznidazole
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Chagas Disease
MeSH Terms: conditions — Chagas Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nifurtimox: Patients treated with Nifurtimox from 1984 to 2017
  Interventions: Other: Clinical Manifestations; Diagnostic Test: Serologic response; Diagnostic Test: Direct method; Behavioral: Adverse events
- Benznidazole: Patients treated with Benznidazole from 1984 to 2017
  Interventions: Other: Clinical Manifestations; Diagnostic Test: Serologic response; Diagnostic Test: Direct method; Behavioral: Adverse events

INTERVENTIONS:
Other: Clinical Manifestations — Clinical manifestations in patients treated with Nifurtimox and Benznidazole
Diagnostic Test: Serologic response — Serologic response in patients treated with Nifurtimox and Benznidazole
Diagnostic Test: Direct method — Direct method tests in patients treated with Nifurtimox and Benznidazole
Behavioral: Adverse events — Adverse events in patients treated with Nifurtimox and Benznidazole

SUMMARY:
Chagas disease is caused by parasite Trypanosoma Cruzi. In Argentina, there is an estimated of 1.600.000 infected people. Due to migration phenomenon, most cases live in urban areas without vectorial transmission.

Pharmacological treatment is given to prevent development of cardiac and gastrointestinal sequelae. There are two available drugs for this disease; Nifurtimox and Benznidazole. They both has proven efficacy for acute face treatment, with different security profiles. There are not enough adequate studies comparing both drugs made in a large number of subjects. Investigators will study 900 patients treated with both drugs and compare security and efficacy in a retrospective cohort.

ELIGIBILITY:
Inclusion Criteria:

- Patients between 0 and 18 years of age with confirmed Chagas disease (defined as patients under 8 months with positive parasitemia or older with 2 positive different techniques for serology) that received treatment with Nifurtimox or Benznidazole.

Exclusion Criteria:

- Patients that abandoned follow-up

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric patients with criteria to receive treatment (Chagas infection confirmed) that received treatment and completed follow-up at Parasitology and Chagas department of Children's Hospital Ricardo Gutierrez, Argentina.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Nifurtimox versus Benznidazole serologic, parasitemia and clinical response for treatment in patients | Patients treated from 1984 to 2017
  To compare Nifurtimox versus Benznidazole treatment efficacy, by measuring serologic response, parasitemia and clinical manifestations in infected patients

SECONDARY OUTCOMES:
Nifurtimox versus Benznidazole security and tolerance | Patients treated from 1984 to 2017
  To compare Nifurtimox versus Benznidazole security profiles, by measuring adverse events in infected patients and comparing both groups (number of adverse reactions, type and severity of reactions)
To compare Chagas disease characteristics associated with treatment | Patients treated from 1984 to 2017
  To describe source of infection, age of acquisition of parasite, diagnosis time frame and clinical manifestations that may be associated with treatment response and compare both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Parasitology and Chagas Service, Buenos Aires Children´s Hospital Ricardo Gutierrez, Buenos Aires, Argentina

REFERENCES:
- [Derived] Falk N, Berenstein AJ, Moscatelli G, Moroni S, Gonzalez N, Ballering G, Freilij H, Altcheh J. Effectiveness of Nifurtimox in the Treatment of Chagas Disease: a Long-Term Retrospective Cohort Study in Children and Adults. Antimicrob Agents Chemother. 2022 May 17;66(5):e0202121. doi: 10.1128/aac.02021-21. Epub 2022 Apr 13. PMID 35416710
- [Derived] Berenstein AJ, Falk N, Moscatelli G, Moroni S, Gonzalez N, Garcia-Bournissen F, Ballering G, Freilij H, Altcheh J. Adverse Events Associated with Nifurtimox Treatment for Chagas Disease in Children and Adults. Antimicrob Agents Chemother. 2021 Jan 20;65(2):e01135-20. doi: 10.1128/AAC.01135-20. Print 2021 Jan 20. PMID 33168612